CLINICAL TRIAL: NCT05708118
Title: Progression of the Ascending Aorta Diameter After Transcatheter Aortic Valve Implantation and Surgical Aortic Valve Replacement in Patients With Bicuspid Aortic Valve.
Brief Title: Progression of Ascending Aorta Diameters in Bicuspid Aortic Valve After Transcatheter or Surgical Replacement.
Acronym: ARDITAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5239
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Bicuspid Aortic Valve; Aortic Valve Stenosis; Aortic Aneurysm; Heart Diseases; Valvular Heart Disease; Valvular Aortic Stenosis; Ascending Aorta Aneurysm
Keywords: Heart valves; Transcatheter aortic valve implantation; Surgical aortic valve replacement; Ascending aorta aneurysm; Bicuspid aortic valve; Bicuspid aortopathy; Transfemoral TAVR
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Valve Stenosis; Aortic Aneurysm; Heart Diseases; Heart Valve Diseases; Aneurysm, Ascending Aorta | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Aortic Valve Replacement (SAVR): Patients who undergo surgical aortic valve replacement through median longitudinal sternotomy.
  Interventions: Diagnostic Test: Echocardiographic assessment.; Diagnostic Test: Computed-tomography assessment
- Transcatheter Aortic Valve Replacement (TAVR): Patients who undergo transcatheter aortic valve replacement through a transfemoral access.
  Interventions: Diagnostic Test: Echocardiographic assessment.; Diagnostic Test: Computed-tomography assessment

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment. — Patients will be contacted to carry out an echocardiography at least 90 days after surgery. Measurements will be taken for aortic annulus, sinuses of Valsalva, sino-tubular junction, tubular ascending aorta. Aortic valve will be assessed as well.
Diagnostic Test: Computed-tomography assessment — All enrolled patients will undergo a multislice CT scan (retrospectively ECG-gated, whenever possible) with standard contrast medium injection protocol of nonionic contrast agent. All post-surgery controls will be performed at least 90 days after surgery. All CT datasets will be analysed on a dedicated workstation for the qualitative and quantitative assessment of the aortic root including measurements for aortic annulus, sinuses of Valsalva, sino-tubular junction, tubular ascending aorta.
  Other Names: CT scan

SUMMARY:
The goal of this prospective, non-randomized, single-center, observational study is to assess whether there is a progressive dilation of ascending aorta after surgical or transcatheter aortic valve replacement (TAVR) in patients who underwent elective aortic valve replacement or TAVR for stenotic bicuspid aortic valve (BAV) at our institution from 2015 to June 2022.

Participants will undergo both a CT and an echocardiographic assessment at least 90 days after surgery.

DETAILED DESCRIPTION:
Bicuspid aortic valve (BAV) is the most common congenital heart defect in adults, affecting 1.3% of the population worldwide. Although valve dysfunction is the most common complication of a bicuspid aortic valve, there is evidence of association of BAV with a specific disease pathology involving the aorta called bicuspid aortopathy. This condition has been proved to predispose to dilatation of all the segments of the proximal aorta both on a genetic and a hemodynamic base, with a reported prevalence of approximately 50% of patients with BAV. Aortic dissection is therefore the most feared complication of BAV aortopathy and BAV itself, but despite a higher relative risk that increases with age, the absolute incidence of aortic dissection remains low.

In elderly population the prevalence of BAV seems to be relatively high as well (incidence of 22% in a reported cohort of octogenarian patients). In the era of transcatheter aortic valve replacement (TAVR), the knowledge of BAV incidence in the elderly is extremely important, assuming that this condition has been considered for years a contraindication to percutaneous procedure by the most. Nevertheless, TAVR has been proved to be a feasible and safe procedure in specific patients deemed at high surgical risk.

As BAV dysfunction tends to reveal earlier than tricuspid ones, when patients are referred to surgery for aortic valve replacement, ascending aorta is often still normal-sized, not deserving surgical treatment, according to current guidelines. It remains controversial whether there is need for concomitant aortic surgery among patients with BAV dysfunction and moderately-dilated aorta, as some authors reported progressive aortic dilatation and aortic dissection even after AVR.

So far, it has never been investigated and there is no information regarding possible differences in the rate of aneurysmal progression in patients with bicuspid aortic valve undergoing surgical or percutaneous aortic valve replacement. A follow-up Computed Tomography (CT) scan is therefore indicated in these patients as chest CT scan is the gold standard for the exact measurement of the aortic diameters.

Aim of this prospective, non-randomized observational study is to assess whether there is a progressive dilation of ascending aorta after surgical or transcatheter aortic valve replacement using CT and echocardiographic imaging in patients with a stenotic BAV who undergo surgical or transcatheter aortic valve replacement.

At the moment no data are available to formulate any hypothesis. Based on our selection criteria a sample size of 150 will be considered in this study, 60% submitted to a surgical approach and 40% to a transcatheter replacement. This sample size is able to detect, in term of effect size, a difference in diameters changes between the 2 procedures from baseline to approximatively 90 days after procedure of about 0.45, considering a significance level of 5% and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bicuspid aortic valve stenosis treated with surgical or transcatheter aortic valve replacement;
* Concomitant ascending aorta aneurysm, with no indication to surgical treatment at the time of intervention;
* Patients with indication to follow-up Chest CT angiography Scan.
* Signed informed consent, inclusive of release of medical information.

Exclusion Criteria:

* Aortic valve replacement in tricuspid valves or bicuspid insufficient valves or endocarditis;
* Aortic valve replacement associated with surgery of ascending aorta/aortic root;
* Aortic valve replacement associated with other cardiac valve surgery;
* Previous cardiac surgery of any kind;
* Patient unable to give informed consent or potentially noncompliant with the study protocol, in the judgment of the investigator;
* Participation in another clinical trial that could interfere with the endpoints of this study;
* Pregnant or breastfeeding at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bicuspid aortic valve stenosis treated with surgical or transcatheter aortic valve replacement and concomitant ascending aorta aneurysm, with no indication to surgical treatment at the time of intervention.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Ascending aorta diameters changes. | At least 90 days after intervention.
  Evaluation of ascending aorta diameters after transcatheter or surgical aortic valve replacement highlighted by both CT and echocardiographic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni A Chiariello, MD, Principal Investigator — Policlinico Agostino Gemelli
Locations (1):
- Policlinico Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verma S, Siu SC. Aortic dilatation in patients with bicuspid aortic valve. N Engl J Med. 2014 May 15;370(20):1920-9. doi: 10.1056/NEJMra1207059. No abstract available. PMID 24827036
- [Background] Michelena HI, Desjardins VA, Avierinos JF, Russo A, Nkomo VT, Sundt TM, Pellikka PA, Tajik AJ, Enriquez-Sarano M. Natural history of asymptomatic patients with normally functioning or minimally dysfunctional bicuspid aortic valve in the community. Circulation. 2008 May 27;117(21):2776-84. doi: 10.1161/CIRCULATIONAHA.107.740878. PMID 18506017
- [Background] Tzemos N, Therrien J, Yip J, Thanassoulis G, Tremblay S, Jamorski MT, Webb GD, Siu SC. Outcomes in adults with bicuspid aortic valves. JAMA. 2008 Sep 17;300(11):1317-25. doi: 10.1001/jama.300.11.1317. PMID 18799444
- [Background] Kim YG, Sun BJ, Park GM, Han S, Kim DH, Song JM, Kang DH, Song JK. Aortopathy and bicuspid aortic valve: haemodynamic burden is main contributor to aortic dilatation. Heart. 2012 Dec;98(24):1822-7. doi: 10.1136/heartjnl-2012-302828. PMID 23204534
- [Background] Fedak PW, Verma S, David TE, Leask RL, Weisel RD, Butany J. Clinical and pathophysiological implications of a bicuspid aortic valve. Circulation. 2002 Aug 20;106(8):900-4. doi: 10.1161/01.cir.0000027905.26586.e8. No abstract available. PMID 12186790
- [Background] Girdauskas E, Borger MA, Secknus MA, Girdauskas G, Kuntze T. Is aortopathy in bicuspid aortic valve disease a congenital defect or a result of abnormal hemodynamics? A critical reappraisal of a one-sided argument. Eur J Cardiothorac Surg. 2011 Jun;39(6):809-14. doi: 10.1016/j.ejcts.2011.01.001. Epub 2011 Feb 20. PMID 21342769
- [Background] Michelena HI, Khanna AD, Mahoney D, Margaryan E, Topilsky Y, Suri RM, Eidem B, Edwards WD, Sundt TM 3rd, Enriquez-Sarano M. Incidence of aortic complications in patients with bicuspid aortic valves. JAMA. 2011 Sep 14;306(10):1104-12. doi: 10.1001/jama.2011.1286. PMID 21917581
- [Background] Roberts WC, Janning KG, Ko JM, Filardo G, Matter GJ. Frequency of congenitally bicuspid aortic valves in patients >/=80 years of age undergoing aortic valve replacement for aortic stenosis (with or without aortic regurgitation) and implications for transcatheter aortic valve implantation. Am J Cardiol. 2012 Jun 1;109(11):1632-6. doi: 10.1016/j.amjcard.2012.01.390. Epub 2012 Mar 27. PMID 22459301
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Vincent F, Ternacle J, Denimal T, Shen M, Redfors B, Delhaye C, Simonato M, Debry N, Verdier B, Shahim B, Pamart T, Spillemaeker H, Schurtz G, Pontana F, Thourani VH, Pibarot P, Van Belle E. Transcatheter Aortic Valve Replacement in Bicuspid Aortic Valve Stenosis. Circulation. 2021 Mar 9;143(10):1043-1061. doi: 10.1161/CIRCULATIONAHA.120.048048. Epub 2021 Mar 8. PMID 33683945
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Yasuda H, Nakatani S, Stugaard M, Tsujita-Kuroda Y, Bando K, Kobayashi J, Yamagishi M, Kitakaze M, Kitamura S, Miyatake K. Failure to prevent progressive dilation of ascending aorta by aortic valve replacement in patients with bicuspid aortic valve: comparison with tricuspid aortic valve. Circulation. 2003 Sep 9;108 Suppl 1:II291-4. doi: 10.1161/01.cir.0000087449.03964.fb. PMID 12970248
- [Background] Girdauskas E, Rouman M, Disha K, Espinoza A, Misfeld M, Borger MA, Kuntze T. Aortic Dissection After Previous Aortic Valve Replacement for Bicuspid Aortic Valve Disease. J Am Coll Cardiol. 2015 Sep 22;66(12):1409-11. doi: 10.1016/j.jacc.2015.07.022. No abstract available. PMID 26383730
- [Background] Burzotta F, Aurigemma C, Romagnoli E, Shoeib O, Russo G, Zambrano A, Verdirosi D, Leone AM, Bruno P, Trani C. A less-invasive totally-endovascular (LITE) technique for trans-femoral transcatheter aortic valve replacement. Catheter Cardiovasc Interv. 2020 Aug;96(2):459-470. doi: 10.1002/ccd.28697. Epub 2020 Jan 11. PMID 31925991
- [Background] Burzotta F, Shoeib O, Aurigemma C, Trani C. Angio-Guidewire-Ultrasound (AGU) Guidance for Femoral Access in Procedures Requiring Large Sheaths. J Invasive Cardiol. 2019 Feb;31(2):E37-E39. doi: 10.25270/jic/18.00173. PMID 30700629